CLINICAL TRIAL: NCT05671874
Title: Pilot Trial of a Web/Mobile/Tablet-based Communication and Goals-of-Care Decision Aid for Clinicians and Families of Severe Acute Brain Injury Patients
Brief Title: Feasibility of a Digital Goals-of-Care Decision Aid for Clinicians and Families of Patients With SABI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Worcester Polytechnic Institute (Other); National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Susanne Muehlschlegel, Professor of Neurology (Neurocritical Care), University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: H00024195; R21NR020231 (NIH)
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hemorrhagic Stroke, Intracerebral; Acute Ischemic Stroke; Traumatic Brain Injury
Keywords: shared decision making; physician-family communication; withdrawal of life sustaining therapies; patient-value congruent care; decision aid; neuroICU; neurocritical care
MeSH Terms: conditions — Hemorrhagic Stroke; Ischemic Stroke; Brain Injuries, Traumatic | interventions — Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: stepped-wedge randomized trial (before-after study)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based Decision Aid + Communication (DA+C) tool (Experimental): Surrogate(s) will read/click through the DA+C tool prior to the clinician-family meeting and complete the integrated worksheet. Surrogate(s) will have unlimited access to the DA+C tool and may return to the tool and edit the worksheet at any time.
  Interventions: Behavioral: Web/mobile/tablet-based digital decision aid + communication (DA+C) tool
- Usual Care (No Intervention): No decision aid

INTERVENTIONS:
Behavioral: Web/mobile/tablet-based digital decision aid + communication (DA+C) tool — The web/mobile/tablet-based digital DA+C toll is designed to enhance communication and shared decision making between clinicians and surrogates of critically ill severe acute brain injury (SABI) with four goals: to 1) prepare families for their surrogate role and discussions with clinicians; 2) provide balanced information to families on prognosis and all available treatment options; 3) provide tailored information about the patient and family to clinicians in advance of family meetings; and 4) serve as a communication guide for clinicians in the clinician-family meeting to facilitate shared decision-making.
  Arms: Web-based Decision Aid + Communication (DA+C) tool

SUMMARY:
The goal is to pilot test a highly accessible, web-based, pragmatic, scalable intervention to overcome ongoing problems with high stakes decision-making by surrogate decision-makers of patients in ICUs with severe acute brain injury (SABI), including those with moderate-severe traumatic brain injury, large hemispheric acute ischemic stroke and intracerebral hemorrhage.

DETAILED DESCRIPTION:
Every 30 seconds an adult in the U.S. suffers a severe acute brain injury (SABI) from traumatic brain injury or large ischemic or hemorrhagic stroke, resulting in 200,000 deaths and >900,000 survivors living with disability annually. Every day, surrogate decision-makers face the difficult "goals of care" decision in intensive care units (ICUs) to continue or withdraw life support while considering the patient's long-term prognosis. In this study, we will pilot test a pragmatic, scalable intervention to overcome ongoing problems with high stakes decision-making by surrogates of patients with SABI in ICUs. These problems are an important target for intervention, because they contribute to 3 major clinical and public health issues: 1) family members struggle in the role of surrogate, leading to lasting symptoms of psychological distress; 2) clinicians are poorly trained in communicating prognosis after SABI, often doing so with variability and bias, inadequately preparing families for their decisions; 3) patients often receive burdensome treatments that they would not choose.

Decision aids improve the quality of patients' decisions based on a large evidence-base, but no empirically validated tools currently exist for surrogate decision-making in SABI patients at high risk for death or disability. This is problematic because surrogates of SABI patients are unprepared for the difficult decisions about the use of life support and patients' potential long-term disability, which hinge on both medical information and the patient's values and preferences. We have developed and refined a tailored digital, web-based decision aid (DA) for families of critically ill SABI patients, conceptually grounded in the Ottawa Decision Support Framework, to enhance, not replace, clinician-family communication. We will leverage a digital platform, which is portable and shareable among family members when geographically distant or not allowed to visit the ICU (as during the COVID-19 pandemic) and allows integration of videos to reach lower-literacy groups. This innovative tool challenges the existing paradigm for decision-making in SABI patients.

This pilot study among 50 surrogates of SABI patients and their clinicians will assess the feasibility of deploying the web-based tool as well as to explore the tools impact on measures of communication and decision-quality.

ELIGIBILITY:
Inclusion criteria for surrogates and patients:

* surrogate is age 18 years or older, no upper age limit;
* documented surrogate decision-maker (official health care proxy, or legal next of kin) of a critically ill severe acute brain injury (SABI) patient ≥ 3 days after admission;
* patient is age 18 years or older, no upper age limit;
* patient has SABI; defined as either traumatic brain injury, spontaneous primary intracerebral hemorrhage (not due to tumor or vascular malformation), or hemispheric acute ischemic stroke;
* patient is"critically ill" defined as either intubated on a mechanical ventilator, or unable to swallow without a feeding tube (even if not intubated/ventilated);
* patient is judged by the attending physician to have ≥40% risk of death or long-term functional impairment, elicited by asking the attending physician, "does this patient have at least a 40% chance of in-hospital mortality or long-term functional impairment?", defined as needing assistance with at least 1 activity of daily living (ADL).
* patient has undergone initial stabilization but remains critically ill;
* surrogate will participate in clinician-family goals of care meeting, either in person or via video- or telephone-conference.
* surrogate must be English speaking and literate

Exclusion Criteria for surrogates and patients:

* devastating patients with severe SABI who die early (within the first 3 days after admission);
* surrogate decision-maker is non-English speaking;
* surrogate decision-maker is illiterate.

Inclusion criteria for clinicians:

* clinical treating attending, or physician trainee (fellow, resident), or licensed affiliated practitioner who will lead the clinician-family meeting when goals-of-care are discussed;
* clinician may decline participation in the outcome measures but cannot restrict the surrogate decision-maker in study participation.

Exclusion criteria for clinicians:

- unwillingness to comply with study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of tool use by surrogate decision-makers | Duration of ICU stay, an expected average of 4 weeks
  Data tracking analytics built into the tool will be employed to determine the extent to which the tools is used as per protocol.
Feasibility of enrolling surrogates in a stepped-wedge (before/after) clinical trial in a neurocritical care setting | Through study completion, estimated 18 months past primary start date
  Measured by meeting target enrollment.
Feasibility of retaining surrogates in a neurocritical care setting | Three-months post SABI
  The number of subjects that complete the long-term follow-up.

SECONDARY OUTCOMES:
Participants' ratings of usability of the tool (Intervention surrogates only) | Duration of ICU stay, an expected average of 4 weeks
  Usability of the tool as measured with the System Usability Scale.
Participants' ratings of perceived effectiveness of the tool in preparing them for decision-making (Intervention surrogates only) | Duration of ICU stay, an expected average of 4 weeks
  Perceived Effectiveness will be measured with an 11-item perceived effectiveness questionnaire using a 5-point Likert scale.
Fidelity to intervention protocol | Through study completion, estimated 18 months past primary start date
  Fidelity to the intervention protocol will be measured using self-checklists by clinicians and review of a random selection of 30% of the audio-recorded clinician-family meetings

OTHER OUTCOMES:
Participants' ratings of what they liked and disliked about the DA+C tool (Intervention surrogates only) | Until right before the scheduled clinician-family meeting, an average of 10-14 days after admission
  Measured by two open ended questions from the Acceptability Scale.
Surrogates' clarity about patient values & preferences | After the scheduled clinician-family meeting, an average of 10-14 days after admission
  We will apply the 3-item Values Clarity Subscale of the Decisional Conflict Scale.
Surrogates' ratings of the degree of shared decision-making | After the scheduled clinician-family meeting, an average of 10-14 days after admission
  We will apply six questions from Quality of Communication Scale pertaining to shared decision-making.
Caregiver Burden | Three-months post SABI
  Measured with the 5-item short form of the Caregiver Burden Scale.
Decision Regret | Three-months post SABI
  Measured using the Decision Regret Scale.
Goals-of-care decision | Hospital discharge up until 3-months post SABI
  Final goals-of-care decision by surrogates (survival vs. withdrawal of life sustaining treatments)
Mortality | Hospital discharge up until 3-months post SABI
  Patient death
Functional status | 3-months post SABI
  We will measure basic activities of daily living with the Glasgow Outcome Scale Extended (GOSE; range 1-8) and the modified Rankin Scale (range 0-6)
Patient-perceived Patient- Centeredness of Care | 3-months post SABI
  To assess patient centeredness of care adapted for use by surrogates

CONTACTS AND LOCATIONS:
Overall Officials: Nils Henninger, MD, PhD, Principal Investigator — University of Massachusetts Chan Medical School; Susanne Muehlschlegel, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - UMass Memorial Hospital, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data not published within the final manuscript will be made available by request from any qualified investigator.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After publication of the main manuscript up until 5 years after publication.
Access Criteria: Requests should be made to the principal investigator smuehlsch[at]jhu.edu

REFERENCES:
- [Background] Muehlschlegel S, Goostrey K, Flahive J, Zhang Q, Pach JJ, Hwang DY. Pilot Randomized Clinical Trial of a Goals-of-Care Decision Aid for Surrogates of Patients With Severe Acute Brain Injury. Neurology. 2022 Oct 3;99(14):e1446-e1455. doi: 10.1212/WNL.0000000000200937. PMID 35853748
- [Background] Goostrey KJ, Lee C, Jones K, Quinn T, Moskowitz J, Pach JJ, Knies AK, Shutter L, Goldberg R, Mazor KM, Hwang DY, Muehlschlegel S. Adapting a Traumatic Brain Injury Goals-of-Care Decision Aid for Critically Ill Patients to Intracerebral Hemorrhage and Hemispheric Acute Ischemic Stroke. Crit Care Explor. 2021 Mar 9;3(3):e0357. doi: 10.1097/CCE.0000000000000357. eCollection 2021 Mar. PMID 33786434
- [Background] Muehlschlegel S, Perman SM, Elmer J, Haggins A, Teixeira Bailey ND, Huang J, Jansky L, Kirchner J, Kasperek-Wynn R, Lipman PD, Yeatts SD, Fetters MD, Dickert NW, Silbergleit R. The Experiences and Needs of Families of Comatose Patients After Cardiac Arrest and Severe Neurotrauma: The Perspectives of National Key Stakeholders During a National Institutes of Health-Funded Workshop. Crit Care Explor. 2022 Mar 4;4(3):e0648. doi: 10.1097/CCE.0000000000000648. eCollection 2022 Mar. PMID 35265851
- [Background] Goostrey K, Muehlschlegel S. Prognostication and shared decision making in neurocritical care. BMJ. 2022 Apr 7;377:e060154. doi: 10.1136/bmj-2021-060154. PMID 35696329
- [Background] Muehlschlegel S, Hwang DY, Flahive J, Quinn T, Lee C, Moskowitz J, Goostrey K, Jones K, Pach JJ, Knies AK, Shutter L, Goldberg R, Mazor KM. Goals-of-care decision aid for critically ill patients with TBI: Development and feasibility testing. Neurology. 2020 Jul 14;95(2):e179-e193. doi: 10.1212/WNL.0000000000009770. Epub 2020 Jun 17. PMID 32554766